CLINICAL TRIAL: NCT04688177
Title: The Association of Cigarette Smoking on Exercise Capacity and Skeletal Muscle Function in Taiwan Adult Smokers
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202010123RIND
Record Dates: First submitted 2020-12-14; First posted 2020-12-29 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2020-12

CONDITIONS: Cigarette Smoking
Keywords: cigarette smoking; exercise capacity; skeletal muscle function; heart rate variability
MeSH Terms: conditions — Cigarette Smoking | interventions — Hand Strength; Respiratory Function Tests; Exercise Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smokers: cigarette smokers male 20 ≤ age ≤ 45 years old female 20 ≤ age ≤ 55 years old
  Interventions: Device: Body Composition; Device: Heart rate variability; Device: Grip Strength; Device: Exhale Carbon Monoxide Concentration; Device: Pulmonary Function Test; Device: Respiratory Muscle Function; Behavioral: Fagerström Test for Nicotine Dependence; Behavioral: Seven-Day Physical Activity Recall Questionnaire; Device: Cardiopulmonary exercise testing
- never smokers: age and gender-matched non-smokers
  Interventions: Device: Body Composition; Device: Heart rate variability; Device: Grip Strength; Device: Exhale Carbon Monoxide Concentration; Device: Pulmonary Function Test; Device: Respiratory Muscle Function; Behavioral: Fagerström Test for Nicotine Dependence; Behavioral: Seven-Day Physical Activity Recall Questionnaire; Device: Cardiopulmonary exercise testing

INTERVENTIONS:
Device: Body Composition — The subjects should lie in the supine position on a non-conducting surface for 5 min. 4 surface electrodes with cables will be attached to the right hand and ankle of subjects.
Device: Heart rate variability — After supine quietly for 20 min, a lead I electrocardiogram will be taken for 5 min.
Device: Grip Strength — The participants will squeeze the hand dynamometer as hard as possible with the dominant hand. 3 successive measurements will be taken.
Device: Exhale Carbon Monoxide Concentration — Subjects in sitting position, performing 1 inspiration, then exhale to carbon monoxide meter.
Device: Pulmonary Function Test — Subjects should be in a sitting position with a nose clip, then perform pulmonary function test. Participants should perform at least 3 acceptable attempts, but no more than 8 attempts in total.
Device: Respiratory Muscle Function — Subject will perform both maximal inspiratory pressure and maximal expiratory pressure for 3 times in sitting position with the nose clip.
Behavioral: Fagerström Test for Nicotine Dependence — Fagerström Test for Nicotine Dependence Traditional Chinese version will be adopted. It is a 6-item questionnaire that could help quantify the smoking frequency, amounts, and level of dependence.
Behavioral: Seven-Day Physical Activity Recall Questionnaire — Physical activity will be measured by the Chinese Version of the Seven-Day Physical Activity Recall Questionnaire. Participants will need to recall the time (hours) they spent in various leisure activities in the past 7 days.
Device: Cardiopulmonary exercise testing — Bruce protocol as the treadmill evaluation protocol will be adopted for cardiopulmonary exercise testing.

SUMMARY:
Background and purpose: Cigarette smoking would post threats to physical health. Even though studies suggested that long-term cigarette smoking would lead to cardiovascular diseases, pulmonary diseases, or even cancer development, the smoking population all around the world was still common. Before progressing into the disease stage, cigarette smokers might have presented decreasing exercise capacity, skeletal muscle function, and cardiac autonomic function as early signs of physiological function decline. The purposes of this study are (1) to investigate the difference in exercise capacity, skeletal muscle function, and cardiac autonomic function between smokers and never smokers, and (2) to test the hypothesis that cigarette smoking is an independent factor associated with exercise capacity.

Methods: This is a cross-sectional observational study. This study will invite 150 participants from community in Taipei City. The body composition will be analyzed by bioelectrical impedance analysis, and resting heart rate variability will be evaluated by the heart rate variability monitor. Besides, grip strength, exhale carbon monoxide concentration, pulmonary function test, respiratory muscle performance will be measured. Moreover, subject will have to fill up the Fagerström Test for Nicotine Dependence and Seven-Day Physical Activity Recall Questionnaire. Last will be the cardiopulmonary exercise testing. Statistical analyses will be performed by statistical software for social sciences (SPSS) statistical package v.21.0 for Windows. (IBM SPSS Statistics for Windows, Version 21.0. Armonk, NY: IBM Corp.) Between-group comparisons of exercise capacity, skeletal muscle function and heart rate variability parameters will be performed using independent Student's t-test. Pearson's correlation coefficient will be used to test the correlations between outcome parameters. Stepwise regression analysis will be used to examine the independent association between smoking and exercise capacity after controlling for confounders. The α level will be set at 0.05. The results of this study would provide the early effects of cigarette smoking on physical function, and highlight the importance of early detection and intervention.

ELIGIBILITY:
Inclusion Criteria:

* male 20 ≤ age ≤ 45 years old
* female 20 ≤ age ≤ 55 years old
* age and gender-matched non-smokers

Exclusion Criteria:

* uncontrolled cardiovascular diseases, neurological diseases, musculoskeletal system problems, or systemic diseases that contraindicate the exercise
* women in pregnancy or menopausal women
* any ongoing medication that has a documented effect on the autonomic nervous system (e.g., tricyclic anti-depressants)
* has been diagnosed with autonomic nervous system disorders

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be invited from community in Taipei City
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | After finishing all the other measurement. The measurement will be lasted 15 minutes.
  Maximal oxygen uptake, VO2max (ml/kg/min), as an indicator of exercise capacity. Cardiopulmonary exercise testing will be used to evaluate the maximal exercise capacity by a computer-controlled breath-by-breath metabolic measurement system (Carefusion Corporation, Yorba Linda, CA, USA) base on the treadmill. Bruce protocol, which is a graded treadmill evaluation protocol will be adopted.

SECONDARY OUTCOMES:
Skeletal muscle function | After finishing heart rate variability and body composition measurement. The measurement will be lasted 5 minutes.
  Skeletal muscle function will be assessed by measuring the grip strength of the dominant hand using a hand dynamometer (Jamar, Jackson, MI, USA).
Cardiac autonomic function | After body composition measurement. The measurement will be lasted 20 minutes.
  Heart rate variability will be measured by HRV monitor (8Z11, Wegene Technology Inc., Taiwan) in this study.
Skeletal muscle mass | After collecting basic data of subjects. The measurement will be lasted 5-10 minutes.
  Skeletal muscle mass (kilogram, kg) will be measured by a bioelectrical impedance analyzer (BIA). (Maltron BioScan 920, Maltron International Ltd., Esgender, UK). The subjects should lie in the supine position on a non-conducting surface for 5 min. Skeletal muscle mass will be calculated by the equation of Janssen and colleagues.
Exhale carbon monoxide concentration | After finishing heart rate variability and body composition measurement. The measurement will be lasted 1-3 minutes.
  Exhale carbon monoxide will be measured by the carbon monoxide meter (CO Check+, MD Diagnostics LTD) for current smoking status evaluation.
Forced expiratory volume in one second | The pulmonary function measurement will be lasted 15 minutes.
  Pulmonary function will be measured by a portable MicroLab® Spirometer (CareFusion, Basingstoke, UK). The outcome measure will include: forced expiratory volume in one second (FEV1, unit: liter).
Forced vital capacity | The pulmonary function measurement will be lasted 15 minutes.
  Pulmonary function will be measured by a portable MicroLab® Spirometer (CareFusion, Basingstoke, UK). The outcome measure will include: forced vital capacity (FVC, unit: liter)
FEV1/FVC ratio | The pulmonary function measurement will be lasted 15 minutes.
  Pulmonary function will be measured by a portable MicroLab® Spirometer (CareFusion, Basingstoke, UK). The outcome measure will include: FEV1/FVC ratio, which is useful for detecting possible dysfunction of the respiratory system in clinical practice.
Respiratory muscle function | After pulmonary function test measurement. The measurement will be lasted 10 minutes.
  Maximal inspiratory pressure (PImax, unit: cmH2O) and maximal expiratory pressure (PEmax, unit: cmH2O) will be measured by a respiratory pressure meter, which could represent the respiratory muscle strength.
Level of nicotine dependence | After respiratory muscle function measurement. The measurement will be lasted 3-5 minutes.
  Fagerström Test for Nicotine Dependence (FTND) Traditional Chinese version will be adopted for quantifying the level of nicotine dependence. FTND is a 6-item questionnaire. The minimum value is 0 points and maximum values is 6 points. The higher score represents the greater nicotine dependence.
Seven-day physical activity recall questionnaire | After respiratory muscle function measurement. The measurement will be lasted 3-5 minutes.
  Physical activity will be measured by the Chinese Version of the Seven-Day Physical Activity Recall Questionnaire. Participants will need to recall the time (hours) they spent in various leisure activities in the past 7 days. The energy expenditure (kcal/day) = metabolic equivalents (METs)*time (hour)*body weight (kg)/7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, College of Medicine, Department of Physical Therapy, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jamal A, Phillips E, Gentzke AS, Homa DM, Babb SD, King BA, Neff LJ. Current Cigarette Smoking Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Jan 19;67(2):53-59. doi: 10.15585/mmwr.mm6702a1. PMID 29346338
- [Background] Chen YL, Wu SC, Chen YT, Hsiao PC, Yu YH, Ting TT, Chen CY, Tu YK, Huang JH, Yang HJ, Li CY, Strong C, Yen CF, Yen CF, Chen WJ. E-Cigarette Use in a Country With Prevalent Tobacco Smoking: A Population-Based Study in Taiwan. J Epidemiol. 2019 Apr 5;29(4):155-163. doi: 10.2188/jea.JE20170300. Epub 2018 Sep 1. PMID 30175730
- [Background] Yoshida T, Tuder RM. Pathobiology of cigarette smoke-induced chronic obstructive pulmonary disease. Physiol Rev. 2007 Jul;87(3):1047-82. doi: 10.1152/physrev.00048.2006. PMID 17615396
- [Background] Tindle HA, Stevenson Duncan M, Greevy RA, Vasan RS, Kundu S, Massion PP, Freiberg MS. Lifetime Smoking History and Risk of Lung Cancer: Results From the Framingham Heart Study. J Natl Cancer Inst. 2018 Nov 1;110(11):1201-1207. doi: 10.1093/jnci/djy041. PMID 29788259
- [Background] Thun MJ, Carter BD, Feskanich D, Freedman ND, Prentice R, Lopez AD, Hartge P, Gapstur SM. 50-year trends in smoking-related mortality in the United States. N Engl J Med. 2013 Jan 24;368(4):351-64. doi: 10.1056/NEJMsa1211127. PMID 23343064
- [Background] Teo KK, Ounpuu S, Hawken S, Pandey MR, Valentin V, Hunt D, Diaz R, Rashed W, Freeman R, Jiang L, Zhang X, Yusuf S; INTERHEART Study Investigators. Tobacco use and risk of myocardial infarction in 52 countries in the INTERHEART study: a case-control study. Lancet. 2006 Aug 19;368(9536):647-58. doi: 10.1016/S0140-6736(06)69249-0. PMID 16920470
- [Background] Watson M, Dardari Z, Kianoush S, Hall ME, DeFilippis AP, Keith RJ, Benjamin EJ, Rodriguez CJ, Bhatnagar A, Lima JA, Butler J, Blaha MJ, Rifai MA. Relation Between Cigarette Smoking and Heart Failure (from the Multiethnic Study of Atherosclerosis). Am J Cardiol. 2019 Jun 15;123(12):1972-1977. doi: 10.1016/j.amjcard.2019.03.015. Epub 2019 Mar 18. PMID 30967285
- [Background] Doll R, Peto R, Boreham J, Sutherland I. Mortality in relation to smoking: 50 years' observations on male British doctors. BMJ. 2004 Jun 26;328(7455):1519. doi: 10.1136/bmj.38142.554479.AE. Epub 2004 Jun 22. PMID 15213107
- [Background] Furlanetto KC, Mantoani LC, Bisca G, Morita AA, Zabatiero J, Proenca M, Kovelis D, Pitta F. Reduction of physical activity in daily life and its determinants in smokers without airflow obstruction. Respirology. 2014 Apr;19(3):369-75. doi: 10.1111/resp.12236. Epub 2014 Feb 2. PMID 24483840
- [Background] Hawari FI. The effect of habitual waterpipe tobacco smoking on pulmonary function and exercise capacity in young healthy males: A pilot study. Respir Med. 2017 Mar;124:102. doi: 10.1016/j.rmed.2017.02.006. Epub 2017 Feb 11. No abstract available. PMID 28237402
- [Background] Mesquita R, Goncalves CG, Hayashi D, Costa Vde S, Teixeira Dde C, de Freitas ER, Felcar JM, Pitta F, Molari M, Probst VS. Smoking status and its relationship with exercise capacity, physical activity in daily life and quality of life in physically independent, elderly individuals. Physiotherapy. 2015 Mar;101(1):55-61. doi: 10.1016/j.physio.2014.04.008. Epub 2014 May 17. PMID 25108641
- [Background] Ben Saad H, Babba M, Boukamcha R, Ghannouchi I, Latiri I, Mezghenni S, Zedini C, Rouatbi S. Investigation of exclusive narghile smokers: deficiency and incapacity measured by spirometry and 6-minute walk test. Respir Care. 2014 Nov;59(11):1696-709. doi: 10.4187/respcare.03058. Epub 2014 Jul 8. PMID 25006270
- [Background] Kobayashi Y, Takeuchi T, Hosoi T, Loeppky JA. Effects of habitual smoking on cardiorespiratory responses to sub-maximal exercise. J Physiol Anthropol Appl Human Sci. 2004 Sep;23(5):163-9. doi: 10.2114/jpa.23.163. PMID 15472461
- [Background] Neves CD, Lacerda AC, Lage VK, Lima LP, Tossige-Gomes R, Fonseca SF, Rocha-Vieira E, Teixeira MM, Mendonca VA. Oxidative stress and skeletal muscle dysfunction are present in healthy smokers. Braz J Med Biol Res. 2016 Oct 24;49(11):e5512. doi: 10.1590/1414-431X20165512. PMID 27783809
- [Background] Morse CI, Wust RC, Jones DA, de Haan A, Degens H. Muscle fatigue resistance during stimulated contractions is reduced in young male smokers. Acta Physiol (Oxf). 2007 Oct;191(2):123-9. doi: 10.1111/j.1748-1716.2007.01721.x. Epub 2007 Jun 5. PMID 17550408
- [Background] Dinas PC, Koutedakis Y, Flouris AD. Effects of active and passive tobacco cigarette smoking on heart rate variability. Int J Cardiol. 2013 Feb 20;163(2):109-15. doi: 10.1016/j.ijcard.2011.10.140. Epub 2011 Nov 17. PMID 22100604
- [Background] McClave AK, Dube SR, Strine TW, Mokdad AH. Associations between health-related quality of life and smoking status among a large sample of U.S. adults. Prev Med. 2009 Feb;48(2):173-9. doi: 10.1016/j.ypmed.2008.11.012. Epub 2008 Dec 6. PMID 19103219
- [Background] Hughes JR, Keely J, Naud S. Shape of the relapse curve and long-term abstinence among untreated smokers. Addiction. 2004 Jan;99(1):29-38. doi: 10.1111/j.1360-0443.2004.00540.x. PMID 14678060
- [Background] Benowitz NL. Nicotine addiction. N Engl J Med. 2010 Jun 17;362(24):2295-303. doi: 10.1056/NEJMra0809890. No abstract available. PMID 20554984
- [Background] Bodner ME, Miller WC, Rhodes RE, Dean E. Smoking cessation and counseling: knowledge and views of Canadian physical therapists. Phys Ther. 2011 Jul;91(7):1051-62. doi: 10.2522/ptj.20100245. Epub 2011 May 5. PMID 21546565
- [Background] Pignataro RM, Ohtake PJ, Swisher A, Dino G. The role of physical therapists in smoking cessation: opportunities for improving treatment outcomes. Phys Ther. 2012 May;92(5):757-66. doi: 10.2522/ptj.20110304. Epub 2012 Jan 6. No abstract available. PMID 22228603
- [Background] Rea BL, Hopp Marshak H, Neish C, Davis N. The role of health promotion in physical therapy in California, New York, and Tennessee. Phys Ther. 2004 Jun;84(6):510-23. PMID 15161417
- [Background] Sung HY, Chang LC, Wen YW, Tsai YW. The costs of smoking and secondhand smoke exposure in Taiwan: a prevalence-based annual cost approach. BMJ Open. 2014 Jul 9;4(7):e005199. doi: 10.1136/bmjopen-2014-005199. PMID 25009135
- [Background] Benowitz NL, Hukkanen J, Jacob P 3rd. Nicotine chemistry, metabolism, kinetics and biomarkers. Handb Exp Pharmacol. 2009;(192):29-60. doi: 10.1007/978-3-540-69248-5_2. PMID 19184645
- [Background] Benowitz NL. Pharmacology of nicotine: addiction, smoking-induced disease, and therapeutics. Annu Rev Pharmacol Toxicol. 2009;49:57-71. doi: 10.1146/annurev.pharmtox.48.113006.094742. PMID 18834313
- [Background] Bierut LJ. Nicotine dependence and genetic variation in the nicotinic receptors. Drug Alcohol Depend. 2009 Oct 1;104 Suppl 1(Suppl 1):S64-9. doi: 10.1016/j.drugalcdep.2009.06.003. Epub 2009 Jul 10. PMID 19596527
- [Background] Kruger K, Dischereit G, Seimetz M, Wilhelm J, Weissmann N, Mooren FC. Time course of cigarette smoke-induced changes of systemic inflammation and muscle structure. Am J Physiol Lung Cell Mol Physiol. 2015 Jul 15;309(2):L119-28. doi: 10.1152/ajplung.00074.2015. Epub 2015 May 22. PMID 26001775
- [Background] Hamari A, Toljamo T, Nieminen P, Kinnula VL. High frequency of chronic cough and sputum production with lowered exercise capacity in young smokers. Ann Med. 2010 Oct;42(7):512-20. doi: 10.3109/07853890.2010.505933. PMID 20662762
- [Background] Rodrigues FM, Loeckx M, Hornikx M, Van Remoortel H, Louvaris Z, Demeyer H, Janssens W, Troosters T. Six years progression of exercise capacity in subjects with mild to moderate airflow obstruction, smoking and never smoking controls. PLoS One. 2018 Dec 26;13(12):e0208841. doi: 10.1371/journal.pone.0208841. eCollection 2018. PMID 30586370
- [Background] Rizzi M, Tarsia P, La Spina T, Cristiano A, Frassanito F, Macaluso C, Airoldi A, Vanni S, Legnani D. A new approach to detect early lung functional impairment in very light smokers. Respir Physiol Neurobiol. 2016 Sep;231:1-6. doi: 10.1016/j.resp.2016.05.010. Epub 2016 May 17. PMID 27224237
- [Background] Rajendra Acharya U, Paul Joseph K, Kannathal N, Lim CM, Suri JS. Heart rate variability: a review. Med Biol Eng Comput. 2006 Dec;44(12):1031-51. doi: 10.1007/s11517-006-0119-0. Epub 2006 Nov 17. PMID 17111118
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Murgia F, Melotti R, Foco L, Gogele M, Meraviglia V, Motta B, Steger A, Toifl M, Sinnecker D, Muller A, Merati G, Schmidt G, Rossini A, Pramstaller PP, Pattaro C. Effects of smoking status, history and intensity on heart rate variability in the general population: The CHRIS study. PLoS One. 2019 Apr 9;14(4):e0215053. doi: 10.1371/journal.pone.0215053. eCollection 2019. PMID 30964923
- [Background] Middlekauff HR, Park J, Moheimani RS. Adverse effects of cigarette and noncigarette smoke exposure on the autonomic nervous system: mechanisms and implications for cardiovascular risk. J Am Coll Cardiol. 2014 Oct 21;64(16):1740-50. doi: 10.1016/j.jacc.2014.06.1201. PMID 25323263
- [Background] Barreiro E, Peinado VI, Galdiz JB, Ferrer E, Marin-Corral J, Sanchez F, Gea J, Barbera JA; ENIGMA in COPD Project. Cigarette smoke-induced oxidative stress: A role in chronic obstructive pulmonary disease skeletal muscle dysfunction. Am J Respir Crit Care Med. 2010 Aug 15;182(4):477-88. doi: 10.1164/rccm.200908-1220OC. Epub 2010 Apr 22. PMID 20413628
- [Background] Kim LJ, Kim N. Difference in lateral abdominal muscle thickness during forceful exhalation in healthy smokers and non-smokers. J Back Musculoskelet Rehabil. 2012;25(4):239-44. doi: 10.3233/BMR-2012-0315. PMID 23220806
- [Background] Saito T, Miyatake N, Sakano N, Oda K, Katayama A, Nishii K, Numata T. Relationship between cigarette smoking and muscle strength in Japanese men. J Prev Med Public Health. 2012 Nov;45(6):381-6. doi: 10.3961/jpmph.2012.45.6.381. Epub 2012 Nov 29. PMID 23230468
- [Background] Tantisuwat A, Thaveeratitham P. Effects of smoking on chest expansion, lung function, and respiratory muscle strength of youths. J Phys Ther Sci. 2014 Feb;26(2):167-70. doi: 10.1589/jpts.26.167. Epub 2014 Feb 28. PMID 24648624
- [Background] Formiga MF, Campos MA, Cahalin LP. Inspiratory Muscle Performance of Former Smokers and Nonsmokers Using the Test of Incremental Respiratory Endurance. Respir Care. 2018 Jan;63(1):86-91. doi: 10.4187/respcare.05716. Epub 2017 Sep 26. PMID 28951469
- [Background] Degens H, Gayan-Ramirez G, van Hees HW. Smoking-induced skeletal muscle dysfunction: from evidence to mechanisms. Am J Respir Crit Care Med. 2015 Mar 15;191(6):620-5. doi: 10.1164/rccm.201410-1830PP. PMID 25581779
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Kemp AH, Quintana DS, Gray MA, Felmingham KL, Brown K, Gatt JM. Impact of depression and antidepressant treatment on heart rate variability: a review and meta-analysis. Biol Psychiatry. 2010 Jun 1;67(11):1067-74. doi: 10.1016/j.biopsych.2009.12.012. Epub 2010 Feb 6. PMID 20138254
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Furlan R, Guzzetti S, Crivellaro W, Dassi S, Tinelli M, Baselli G, Cerutti S, Lombardi F, Pagani M, Malliani A. Continuous 24-hour assessment of the neural regulation of systemic arterial pressure and RR variabilities in ambulant subjects. Circulation. 1990 Feb;81(2):537-47. doi: 10.1161/01.cir.81.2.537. PMID 2297860
- [Background] Tengvall M, Ellegard L, Malmros V, Bosaeus N, Lissner L, Bosaeus I. Body composition in the elderly: reference values and bioelectrical impedance spectroscopy to predict total body skeletal muscle mass. Clin Nutr. 2009 Feb;28(1):52-8. doi: 10.1016/j.clnu.2008.10.005. Epub 2008 Nov 17. PMID 19010572
- [Background] Janssen I, Heymsfield SB, Baumgartner RN, Ross R. Estimation of skeletal muscle mass by bioelectrical impedance analysis. J Appl Physiol (1985). 2000 Aug;89(2):465-71. doi: 10.1152/jappl.2000.89.2.465. PMID 10926627
- [Background] Chien MY, Huang TY, Wu YT. Prevalence of sarcopenia estimated using a bioelectrical impedance analysis prediction equation in community-dwelling elderly people in Taiwan. J Am Geriatr Soc. 2008 Sep;56(9):1710-5. doi: 10.1111/j.1532-5415.2008.01854.x. Epub 2008 Aug 6. PMID 18691288
- [Background] Hamilton A, Balnave R, Adams R. Grip strength testing reliability. J Hand Ther. 1994 Jul-Sep;7(3):163-70. doi: 10.1016/s0894-1130(12)80058-5. PMID 7951708
- [Background] Marrone GF, Paulpillai M, Evans RJ, Singleton EG, Heishman SJ. Breath carbon monoxide and semiquantitative saliva cotinine as biomarkers for smoking. Hum Psychopharmacol. 2010 Jan;25(1):80-3. doi: 10.1002/hup.1078. PMID 19998321
- [Background] Cheng S, Lyass A, Massaro JM, O'Connor GT, Keaney JF Jr, Vasan RS. Exhaled carbon monoxide and risk of metabolic syndrome and cardiovascular disease in the community. Circulation. 2010 Oct 12;122(15):1470-7. doi: 10.1161/CIRCULATIONAHA.110.941013. Epub 2010 Sep 27. PMID 20876437
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Payne TJ, Smith PO, McCracken LM, McSherry WC, Antony MM. Assessing nicotine dependence: a comparison of the Fagerstrom Tolerance Questionnaire (FTQ) with the Fagerstrom Test for Nicotine Dependence (FTND) in a clinical sample. Addict Behav. 1994 May-Jun;19(3):307-17. doi: 10.1016/0306-4603(94)90032-9. PMID 7942248
- [Background] Fagerstrom KO. Measuring degree of physical dependence to tobacco smoking with reference to individualization of treatment. Addict Behav. 1978;3(3-4):235-41. doi: 10.1016/0306-4603(78)90024-2. No abstract available. PMID 735910
- [Background] Huang CL, Lin HH, Wang HH. Evaluating screening performances of the Fagerstrom tolerance questionnaire, the Fagerstrom test for nicotine dependence and the heavy smoking index among Taiwanese male smokers. J Clin Nurs. 2008 Apr;17(7):884-90. doi: 10.1111/j.1365-2702.2007.02054.x. PMID 18321287
- [Background] Gross LD, Sallis JF, Buono MJ, Roby JJ, Nelson JA. Reliability of interviewers using the Seven-Day Physical Activity Recall. Res Q Exerc Sport. 1990 Dec;61(4):321-5. doi: 10.1080/02701367.1990.10607494. PMID 2132889
- See also: Health Promotion Administration, Ministry of Health and Welfare, Taiwan. Taiwan Tobacco Control Annual Report 2015. 2015. — https://www.hpa.gov.tw/Pages/Detail.aspx?nodeid=1054&pid=6010
- See also: Liu JY, Chen TJ, Hwang SJ. Predicting Factors of Smoking Cessation in Outpatient Smoking Cessation Clinic. Taiwan J Fam Med 2017; 27: 146-153. — https://www.tafm.org.tw/ehc-tafm/s/viewDocument?documentId=4d29bb25941b459fa89f45a3aeff1ad5
- See also: Tsai YM. The Effect of Smoking on the Recuperation after Exercise. Journal of Exercise Physiology and Fitness, (3), 2005. — https://www.airitilibrary.com/Publication/alDetailedMesh?docid=1815638x-200512-x-3-31-38-a
- See also: Chung CY, Hung CC, Hwang SJ, Chen HC. The Application of Bioimpedance Analysis in Internal Medicine. J Intern Med Taiwan 2012; 23: 245-253. — https://www.airitilibrary.com/Publication/alDetailedMesh?DocID=10167390-201208-201210020010-201210020010-245-253
- See also: 衛生福利部國民健康署健康九九網站。尼古丁成癮度量表。2020。Access date: 2020/07/28. — https://health99.hpa.gov.tw/onlineQuiz/smoking
- See also: Chien MY, Wu TY, Kwan WK, Chien CL. Reliability of the Chinese Version of the 7-day Recall Physical Activity Questionnaire and Its Correlation with Impairments of Disease and Function. FJPT 2003; 28(1):01-08. — https://www.airitilibrary.com/Publication/alDetailedMesh?DocID=15632555-200302-28-1-1-8-a